CLINICAL TRIAL: NCT02432560
Title: Multicenter International Durability and Safety of Sirolimus in LAM Trial (MIDAS)
Brief Title: Safety and Durability of Sirolimus for Treatment of LAM
Acronym: MIDAS
Status: Recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); The LAM Foundation (Other)
Responsible Party: Principal Investigator, Francis McCormack, Professor, University of Cincinnati
Other Study IDs: MIDAS; 1U54HL127672 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-05-04 (Estimated); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Lymphangioleiomyomatosis; LAM; rare lung; Rare Lung Disease
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Sirolimus; Everolimus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Everolimus: women over age 18 who have LAM and are currently taking, have previously failed or been intolerant of, or who are considering taking everolimus as part of their clinical care
  Interventions: Drug: Everolimus
- Sirolimus: women over age 18 who have LAM and are currently taking, have previously failed or been intolerant of, or who are considering taking sirolimus as part of their clinical care
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus treatment will be part of a participant's clinical care and will be managed by their physician.
  Other Names: Rapamune, rapamycin
  Groups: Sirolimus
Drug: Everolimus — Everolimus treatment will be part of a participant's clinical care and will be managed by their physician.
  Other Names: Afinitor
  Groups: Everolimus

SUMMARY:
The MIDAS study aims to follow male and female LAM patients who are currently taking, have previously failed or been intolerant of, or may (at some time in the future) take mTOR inhibitors (sirolimus or everolimus) as part of their clinical care. Adult female TSC patients may also enroll, with or without lung cysts.

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis (LAM) is an uncommon disease affecting women. It is associated with cystic lung destruction and progressive respiratory failure. The Multicenter International LAM Efficacy of Sirolimus (MILES) Trial, led by the investigators' research team, demonstrated that mTOR (mammalian target of rapamycin) inhibition with sirolimus was an effective therapy that stabilized decline in FEV1 (forced expiratory volume). However, lung function decline resumed when the drug was stopped at the one year point in MILES, suggesting that therapy is suppressive rather than remission-inducing, and may need to be lifelong. There is therefore a need to understand whether long-term therapy with sirolimus is safe and effective. To accomplish this goal, the investigators will conduct the Multicenter International Durability and Safety of Sirolimus in LAM Trial (MIDAS). This is an observational, real world registry. The investigators propose to enroll 600 LAM patients who are on, have previously failed or been intolerant of or are considering taking sirolimus or everolimus for clinical reasons in a longitudinal observational study. This registry will follow lung function tests and adverse events that are obtained for clinical purposes over periods of at least 2 years. The decision to treat with mTOR inhibitor therapy is made by the clinician and the patient, and will be managed by the participant's clinician. This study will help us to refine treatment for patients with LAM and determine if long term suppressive therapy with sirolimus can prevent progression to later stages of disease. This research will be accomplished as part of the NIH/NCATS Rare Lung Disease Consortium, with data stored and analyzed by the Database Management Coordinating Center (DMCC) at the University of South Florida.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, age 18 or over
* Diagnosis of LAM based on ATS/JRS criteria
* Signed and dated informed consent
* On chronic therapy, newly treated or may be considered for therapy with mTOR inhibitors or previously intolerant of or having failed mTOR inhibitor therapy

Exclusion Criteria:

* Inability to attend at least one RLD Clinic visit per year
* Inability to give informed consent
* Inability or unwillingness to perform pulmonary function testing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rare Lung Disease Clinical Network Consortium Clinics
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Long term safety of mTOR inhibitor treatment in LAM | 2-5 years
  Symptoms and adverse events will be recorded
Efficacy - FEV1 slope | 2-5 years
  Rate of change in FEV1 in ml/month
Efficacy -10% reduction in FEV1 | 2-5 years
  time from enrollment to 10% or greater reduction in FEV1(forced expiratory volume) in months

SECONDARY OUTCOMES:
Effect of long term sirolimus on quality of life | 2-5 years
  Evaluate ATAQ-LAM QOL responses over time

CONTACTS AND LOCATIONS:
Overall Officials: Francis X McCormack, MD, Study Director — University of Cincinnati
Locations (20):
- United States (20):
  - Stanford University Medical Center, Stanford, California
  - National Jewish Health, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Loyola University Medical Center, Chicago, Maywood, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Center, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington